CLINICAL TRIAL: NCT05818826
Title: Composite Adverse Events Compared Early Versus Conventional Cessation of Hydrocortisone in Patients With Septic Shock: Randomized-controlled Trial
Brief Title: Early Versus Conventional Cessation of Hydrocortisone in Septic Shock
Acronym: CESSHYDRO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SI 012/2023
Record Dates: First submitted 2023-03-19; First posted 2023-04-19 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Septic Shock; Adverse Event; Hydrocortisone; Hyperglycemia; Hypernatremia; Muscle Weakness; Superimposed Infection
Keywords: septic shock; composite adverse events; hydrocortisone; hyperglycemia; hypernatremia; muscle weakness; superimposed infection
MeSH Terms: conditions — Shock, Septic; Hyperglycemia; Hypernatremia; Muscle Weakness; Superinfection | interventions — Saline Solution; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Pharmacist who does not involve in patient enrollment nor treatment will prepared hydrocortisone or placebo in the identical container, before the study drug will be discontinued from patients , according to their treatment arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- early cessation group (Experimental): The pharmacist uses 100 ml of normal saline solution, packed out in the same format, dose, and administration of the drug were exactly the same as in the conventional cessation group. The experimental starts after required dose of vasopressor less than 0.1 mcg/kg/min. The nurse serially records capillary blood glucose and serum sodium following the doctor's order.
  Interventions: Drug: normal saline solution
- conventional cessation group (Placebo Comparator): The pharmacist prepared hydrocortisone and normal saline solution 100 ml starts dose at least 200 mg/day according to doctor's order after patient meets the criteria of refractory septic shock then continues conventional cessation of hydrocortisone according to doctor's order after required dose of vasopressor less than 0.1 mcg/kg/min. The nurse serially records capillary blood glucose and serum sodium following the doctor's order.
  Interventions: Drug: Hydrocortisone and normal saline solution

INTERVENTIONS:
Drug: normal saline solution — Prepare 100 ml of normal saline solution, packed out in the same format, dose, and administration of the drug were exactly the same as in the conventional cessation group.
  Other Names: early cessation group
  Arms: early cessation group
Drug: Hydrocortisone and normal saline solution — Prepare hydrocortisone with normal saline solution 100 ml starts dose at least 200 mg/day according to doctor's order after patient meets the criteria of refractory septic shock then continues conventional cessation of hydrocortisone according to doctor's order after required dose of vasopressor less than 0.1 mcg/kg/min.
  Other Names: conventional cessation group
  Arms: conventional cessation group

SUMMARY:
Septic shock is one of the causes of death in ICU and hospital. Refractory shock is the problem which healthcare providers should recognize though it is difficult to handle with. The corticosteroid called hydrocortisone is one of the treatment in refractory septic shock which requires vasopressor to maintain blood pressure. In recovery phase of septic shock and weaning off vasopressor, there is no definite way to taper off hydrocortisone.

DETAILED DESCRIPTION:
According to secondary outcomes of several studies analyzed in systemic review was shown adverse events from corticosteroid uses including hyperglycemia, hypernatremia, muscle weakness, and superimposed infection. This trials will compare composite adverse events in early versus conventional cessation of hydrocortisone in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patient >= 18 years old
* Diagnosis Septic shock from the definition of SEPSIS III criteria in intensive care unit or medicine ward or surgical ward at Siriraj hospital
* Received at least 1 catecholamines and hydrocortisone at least 200 mg/d
* Maintain mean arterial pressure >= 65 mmHg even if titrate down catecholamines until low dose (<=0.1 mcg/kg/min)

Exclusion Criteria:

* Patient sign Do not resuscitation and terminally ill
* Pregnancy
* Need long term steroid use due to other medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Composite adverse events of early versus conventional cessation of hydrocortisone | within 14 days after randomization or until discharge from hospital, whichever came first
  including level of capillary blood glucose >= 180mg/dL(Hyperglycemia) , Plasma level of sodium>= 150mmol/L(Hypernatremia), new onset of infection , and neuromuscular weakness(muscular impairment rating scale>1

SECONDARY OUTCOMES:
Number of participants with 28-day mortality from any cause or until discharge from hospital | 28-day mortality from any cause start until 28 day after randomization or until discharge from hospital, whichever came first
  death from any cause until 28-day after randomization or until discharge from hospital
Concentration of insulin needed due to hyperglycemia | within 14 days after randomization or until discharge from hospital, whichever came first
  Total insulin used to lower capillary blood sugar if level of glucose more than 180 mg/dL
Number of participants with hypoglycemia | within 14 days after randomization or until discharge from hospital, whichever came first
  Number of participants with capillary blood glucose < 80 mg/dL
Number of participants with capillary blood glucose ≥ 150 mg/dL | within 14 days after randomization or until discharge from hospital, whichever came first
  Number of participants with capillary blood glucose ≥ 150 mg/dL
Time of vasopressor reinitiation until 14 day after randomization or until hospital discharge | within 14 days after randomization or until discharge from hospital, whichever came first
  Duration measured as hours from off vasopressor until re-initiation at least 0.05 mcg/kg/min until 14 day after randomization or until hospital discharge
Time to need of fluid bolus | within 14 days after randomization or until discharge from hospital, whichever came first
  Duration measured as hours from randomization until fluid bolus at least 250 ml in 10-15 minutes until 14 day after randomization or until hospital discharge
Time to reversal of shock | within 14 days after first dose of hydrocortisone or until discharge from hospital, whichever came first
  Duration measured as hours from randomization until off vasopressor
Number of participants with New onset of infection within 28 days | 28 days
  Number of participants with New onset of infection within 28 days
Duration of ICU length of stay | 14 days after first dose hydrocortisone or until discharge from hospital, whichever came first
  Duration measured as days from randomization until discharge from ICU
Duration of Ventilator free day | 14 days after first dose hydrocortisone or until discharge from hospital, whichever came first
  Duration measured as hours from off ventilator until on ventilator or reintubation
Number of participants with Lung injury score at day 1, day 3, day 7 after first dose hydrocortisone | 7 days after randomization or until discharge from hospital, whichever came first
  Number of participants with Lung injury score at day1, day3, day7 after first dose hydrocortisone
Level of minimum and maximum mean arterial pressure | within 14 days after randomization or until discharge from hospital, whichever came first
  Level of minimum and maximum mean arterial pressure until 14 days after randomization or until hospital discharge
Number of participants with Alive days in 28 days with free mechanical ventilator | 28 days after randomization or until discharge from hospital, whichever came first
  Number of participants who survive in 28 days with free mechanical ventilator
Number of participants with Alive days in 28 days with free renal replacement therapy | 28 days after randomization or until discharge from hospital, whichever came first
  Number of participants who survive in 28 days with free mechanical ventilator
Number of participants with Alive days in 28 days with free organ supports | 28 days after randomization or until discharge from hospital, whichever came first
  Number of participants who survive in 28 days with free mechanical ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Surat Tongyoo, Doctor, Principal Investigator — Mahidol University
Locations (1):
- Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Anonymous identification data will be prepared per request, after study publication 6 months
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 6 months post study publication
Access Criteria: Request to principal investigation, after protocol approval from ethical committee